CLINICAL TRIAL: NCT07271680
Title: The Effect of Smartphone Addiction to Uterine Artery Blood Flow, Fetal Heart Rate, and Fetal Birth Weight in the Third Trimester of Pregnancy
Brief Title: Effects of Smartphone Addiction to Fetal Parameters in Pregnancy
Acronym: ESAFPP
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Antalya City/ Anatolian Hospit
Record Dates: First submitted 2025-09-04; First posted 2025-12-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Smart Phone Addiction
Keywords: pregnancy; uterine blood flow; fetal heart rate; birth weight; smart phone addiction
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with smartphone addiction: According to Smartphone Addiction Scale - Short Version (SAS-SV) pregnant women with a score of 33 or higher (accepted as addicted to their smartphones according to the scale).
- Pregnant women without smartphone addiction: According to SAS-SV pregnant women with a score of 32 or lower (accepted as not addicted to their smartphones according to the scale).

SUMMARY:
This prospective cohort study investigates the relationship between smartphone addiction and fetal health parameters at the third trimester of pregnancy. Pregnant women will be evaluated for smartphone addiction, and fetal heart rate, uterine artery blood flow indices (Resistive Index, Systolic/Diastolic ratio), and birth weight will be measured. The hypothesis is that smartphone addiction may negatively affect fetal outcomes, leading to higher fetal heart rate, impaired uterine artery blood flow, and lower birth weight.

Although no direct studies have examined smartphone addiction and these fetal parameters together, related evidence suggests possible adverse effects of mobile phone exposure on oxidative stress, infant birth weight, fetal heart rate variability, and anthropometric measures. This study is among the first to specifically link smartphone addiction with maternal-fetal outcomes, offering new insights into environmental risk factors during late pregnancy. The findings aim to provide healthcare professionals with evidence based guidance for counseling pregnant women on safe smartphone use to protect maternal and fetal health.

DETAILED DESCRIPTION:
The Relationship of Smartphone Addiction to Fetal Heart Rate, Fetal Birth Weight, and Uterine Artery Blood Flow in the Third Trimester of Pregnancy This is a prospective cohort study. Fetal heart rate, uterine artery blood flow, and infant birth weight will be measured during the third trimester (28 weeks and beyond) of pregnancy to examine the relationship between these values and smartphone addiction.

Smartphone use is increasingly common today, and the potential effects of this on maternal and fetal health, especially during pregnancy, are becoming an important research topic. The third trimester of pregnancy is a critical period of rapid growth and preparation for birth, and investigating the effects of exposure to environmental factors on the fetus during this period is of great importance. This study aims to make a significant contribution to the literature by examining the potential effects of smartphone addiction on fetal heart rate, uterine artery blood flow parameters, and birth weight during the third trimester of pregnancy. H1: In pregnant women with smartphone addiction in the third trimester, fetal health parameters will be impaired. Fetal heart rate values will be negatively affected (higher). Uterine artery blood flow indicators will be impaired (increased Resistive Index (RI) and Systolic/Diastolic (S/D) ratio). Birth weight will be lower.

H0: There will be no statistically significant difference in fetal health parameters (fetal heart rate, uterine artery RI, S/D ratio, birth weight) between pregnant women with smartphone addiction and those without addiction.

There is no direct study on the specific relationship between smartphone addiction or screen time in the last trimester of pregnancy and fetal heart rate, uterine artery blood flow, and birth weight. However, related research themes exist:

A study conducted in Turkey demonstrated that mobile phone exposure during pregnancy has the potential to cause oxidative stress by increasing oxidant levels and decreasing antioxidant levels in cord blood (1). A study conducted in Japan found that excessive phone use was associated with lower average birth weight and a higher incidence of emergency baby transport (2). A systemic review showed that electromagnetic field radiation exposure was associated with hormonal, thermal, and cardiovascular changes among adults. Only four of the reviewed studies were conducted among pregnant women. These studies reported that radiation exposure during pregnancy was associated with miscarriages, fluctuations in fetal temperature and heart rate variability, as well as infant anthropometric measurements (3).

This study makes a unique contribution to the literature because it is one of the first to examine the impact of smartphone addiction on fetal heart rate, uterine artery blood flow, and the risk of low birth weight. While existing research generally focuses on the general effects of mobile phone use, this study provides a more comprehensive analysis by assessing the level of addiction. Furthermore, the use of an objective measure such as fetal heart rate enhances the scientific value of the study.

The primary objective of this study was to determine the potential effects of smartphone addiction during the last trimester of pregnancy on fetal health indicators and low birth weight. This will contribute to the development of more informed recommendations for smartphone use during pregnancy and the protection of maternal and fetal health. The resulting data will provide healthcare professionals with a scientific basis for better counseling pregnant women.

Statistical analysis clarification:

Although participants were initially planned to be compared according to the established clinical cut-off of the Smartphone Addiction Scale-Short Version (SAS-SV ≥33 vs <33), the observed distribution resulted in a relatively small number of participants meeting the addiction threshold. Therefore, the primary statistical analyses were conducted using the total SAS-SV score as a continuous variable to preserve information and optimize statistical power. Comparisons based on the clinical addiction cut-off were performed as secondary and sensitivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of singleton pregnancy
* Must be in the third trimester of pregnancy (confirmed by ultrasound)
* Must agree to participate voluntarily in the study and signing the informed consent form
* Must own a smartphone

Exclusion Criteria:

* Clinical diagnosis of multiple pregnancy
* History of miscarriage in previous pregnancies (3 or more)
* Clinical diagnosis of chronic systemic diseases (e.g., diabetes, hypertension, thyroid disease)
* Clinical diagnosis of fetal anomaly in the fetus
* Drug or substance addiction
* Clinical diagnosis of serious psychiatric disorder
* Cigarette smoker

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of pregnant women in their third trimester (34-36 weeks of gestation) who present to Obstetric Clinics for routine antenatal follow-up. Eligible participants are biological females, aged 18-40 years, with singleton pregnancies, smartphone users, and without chronic systemic disease, fetal anomalies, or other exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Fetal Heart Rate Measurement | At baseline visit (single ultrasound assessment on the day of enrollment)
  Fetal heart rate will be measured using ultrasound. Measurements will be performed by an experienced obstetrician and gynecologist in accordance with standard protocols.
Resistance Index Measurement | At baseline visit (single Doppler assessment on the day of enrollment)
  RI will be checked and noted. obtained data will be compared with reference data for the given gestational age, and uterine blood flow will be coded as 0 for decreased and 1 for normal.
Systolic/ Diastolic Ratio Measurement | At baseline visit (single Doppler assessment on the day of enrollment)
  S/D ratio will be checked and noted. The obtained data will be compared with reference data for the given gestational age, and uterine blood flow will be coded as 0 for decreased and 1 for normal.

SECONDARY OUTCOMES:
Birth weight measurement | At delivery (from enrollment until birth, assessed once at the time of delivery, up to approximately 12 weeks after enrollment)
  The baby's initial weight, measured on a newborn scale in the delivery room, will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Selkin Yilmaz Muluk, MD, Study Director — Ministry of Health Antalya City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Ministry of Health Antalya City Hospital, Antalya
  - Antalya Anatolia Hospital, Antalya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to researchers who provide a methodologically sound and ethically approved research proposal. Data will be shared via a secure, designated platform, and a data use agreement will be required to ensure compliance with privacy and ethical standards.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years
Access Criteria: De-identified individual participant data will be made available to researchers who provide a methodologically sound and ethically approved research proposal. Data will be shared via a secure, designated platform, and a data use agreement will be required to ensure compliance with privacy and ethical standards.
URL: https://zenodo.org/records/16931249

REFERENCES:
- [Background] Cirak Y, Yilmaz GD, Demir YP, Dalkilinc M, Yaman S. Pregnancy physical activity questionnaire (PPAQ): reliability and validity of Turkish version. J Phys Ther Sci. 2015 Dec;27(12):3703-9. doi: 10.1589/jpts.27.3703. Epub 2015 Dec 28. PMID 26834336
- [Background] Park S, Marcotte R, Staudenmayer J, Sirard J, VanKim N, Pekow P, Strath S, Freedson P, Chasan-Taber L. Validity of the Pregnancy Physical Activity Questionnaire Short Form (PPAQ-SF). Am J Epidemiol. 2024 Oct 2:kwae382. doi: 10.1093/aje/kwae382. Online ahead of print. PMID 39359005
- [Background] Evren C, Dalbudak E, Topcu M, Kutlu N, Evren B, Pontes HM. Psychometric validation of the Turkish nine-item Internet Gaming Disorder Scale-Short Form (IGDS9-SF). Psychiatry Res. 2018 Jul;265:349-354. doi: 10.1016/j.psychres.2018.05.002. Epub 2018 May 4. PMID 29793049
- [Background] Kwon M, Kim DJ, Cho H, Yang S. The smartphone addiction scale: development and validation of a short version for adolescents. PLoS One. 2013 Dec 31;8(12):e83558. doi: 10.1371/journal.pone.0083558. eCollection 2013. PMID 24391787
- [Background] Lu X, Oda M, Ohba T, Mitsubuchi H, Masuda S, Katoh T. Association of excessive mobile phone use during pregnancy with birth weight: an adjunct study in Kumamoto of Japan Environment and Children's Study. Environ Health Prev Med. 2017 Jun 8;22(1):52. doi: 10.1186/s12199-017-0656-1. PMID 29165149
- [Background] Özen G, Kahvecioğlu D, Bulut İ, Erel Ö, Neşelioğlu S, Üstün Y, Taşar MA. Effect of Mobile Phone Usage During Pregnancy on Total Oxidant and Antioxidant Levels in Cord Blood. J Behcet Uz Child Hosp 2023;13(3):177-184.